CLINICAL TRIAL: NCT04517591
Title: Reducing Sedentary Time in Post-bariatric Patients: The Take a STAND for Health Study
Brief Title: Reducing Sedentary Time in Bariatric: The Take a STAND for Health Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26581219.6.0000.0068
Record Dates: First submitted 2020-08-12; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Obesity, Morbid; Bariatric Surgery
MeSH Terms: conditions — Obesity, Morbid | interventions — Health

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Take a STAND for health (Experimental): A newly developed personalized intervention focused on replacing sedentary time with light-(or very light-) intensity physical activity
  Interventions: Behavioral: The Take a STAND for health
- Control (No Intervention): The control group will receive all regular medical care and advice on healthy lifestyle including the promotion of recommended physical activity levels and health nutrition.

INTERVENTIONS:
Behavioral: The Take a STAND for health — A 4-month parallel-group randomised controlled trial will be performed, in which patients post-bariatric surgery will be assessed at baseline pre-surgery (PRE-BAR), 3 months after surgery and pre-intervention (PRE-INT) and 4 months after intervention (POST). Moreover, a sub-sample of patients will perform a randomised crossover trial at baseline (PRE). Patients will complete three experimental sessions in a random manner, as follows: Prolonged sitting (SIT), in which participants engaged in prolonged sitting throughout an 5-h period and were instructed to minimize excessive movement; Exercise followed by prolonged sitting (EX), in which participants performed a 30-min moderate-to-vigorous exercise bout on a treadmill, subsequently, participants engaged in prolonged sitting as described for SIT; Light-intensity breaks (BR), in which participants completed a 3-min bout of light-intensity walking every 30 min of sitting throughout the experimental period.
  Arms: Take a STAND for health

SUMMARY:
This research program aims to comprehensively investigate the clinical, physiological, metabolic, and molecular effects of reducing sedentary behavior in post-bariatric patients. To this aim, we will conduct a crossover trial and a randomized controlled trial. The crossover trial aims to unravel potential mechanisms underlying the metabolic, physiological and molecular effects of breaking up sedentary time with light-intensity physical activity versus carrying out the minimum amount of daily exercise at once and then remaining sedentary versus simply remaining sedentary throughout all sessions, in a well-controlled laboratorial condition. The 4-month parallel-group randomized controlled trials aim to investigate the feasibility and efficacy of a newly developed personalized intervention focused on replacing sedentary time with light- (or very light-) intensity physical activity in these patients. A multitude of gold-standard techniques will be applied to evaluate the effects of the intervention on several outcomes, including sedentary time (primary outcome), physical activity levels, clinical parameters specific to each condition, cardiometabolic risk factors, immune function, and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria: Women aged 20 to 50 years with BMI ≥ 35 kg / m2 and associated comorbidities, or BMI ≥ 40 kg / m2 who are about to undergo Roux-en-Y gastric bypass surgery at the Metabolic and Bariatric Surgery Unit of the Faculty of Medicine.

-

Exclusion Criteria: Exclusion criteria will involve sedentary time (sitting / reclining) <8 hours per day; anemia; hypothyroidism; current malignancy or history of cancer within the past 5 years; cardiovascular disease; neurological disorders; any physical disabilities that could hamper physical testing; and being physically active (i.e., participation in ≥ 150 minutes per week of moderate-to-vigorous physical activity in bouts of ≥ 10 minutes, or ≥ 75 minutes per week of vigorous-intensity physical activity).

-

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-07 (Estimated); Primary Completion 2022-10-08 (Estimated); Study Completion 2022-10-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to follow-up on sedentary behaviour | 4 months
  Sedentary behaviour will be assessed by ActivPAL™

SECONDARY OUTCOMES:
Change from baseline to follow-up on physical activity levels | 4 months
  Physical activity levels will be assessed by ActiGraph GT3X®
Change from baseline to follow-up on body composition | 4 months
  Lean mass, fat mass and bone mass will be assessed by densitometry (DEXA)
Change from baseline to follow-up on aerobic capacity | 4 months
  Aerobic capacity will be assessed by a maximal cardiopulmonary exercise test
Change from baseline to follow-up on food intake | 4 months
  Food intake will be assessed by means of three 24-hours food recalls
Change from baseline to follow-up on office and ambulatory blood pressure | 4 months (RCT) and 5 hours (crossover)
  Office and ambulatory blood pressure will be assessed by automated devices
Change from baseline to follow-up on quality of life | 4 months
  Quality of life will be assessed by Bariatric Analysis and Reporting Outcome questionnaire
Change from baseline to follow-up on functional capacity and fatigue | 4 months
  Functional capacity will be assessed by Timed Up-And-Go, Time-Stands and handgrip tests. Fatigue will be assessed by fatigue severity scale and Chalder fatigue scale.
Change from baseline to follow-up on cardiovascular risk score | 4 months
  Cardiovascular risk score will be assessed by Framingham score
Change from baseline to follow-up on sleep apnea | 4 months
  Sleep apnea will be assessed by polysomnography
Change from baseline to follow-up on autonomic function | 4 months
  Autonomic function will be assessed by heart rate variability
Change from baseline to follow-up on cardiovascular and respiratory chemoreflex control | 4 months
  Cardiovascular and respiratory chemoreflex control will be assessed by hyperoxia and hypoxia protocol

OTHER OUTCOMES:
Change from baseline to follow-up on vascular function | 4 months (RCT) and 5 hours (crossover)
  Vascular function will be assessed by flow-mediated dilatation
Change from baseline to follow-up on blood markers | 4 months (RCT) and 5 hours (crossover)
  Insulin sensitivity: fasting glucose and insulin; Lipid profile: Total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides
Change from baseline to follow-up on inflammatory markers | 4 months
  Pro- and anti-inflammatory cytokines: IL-1, IL-1ra, IL-6, IL-10 e TNF-alpha;
Change from baseline to follow-up on oral glucose tolerance test | 4 months
  Assessed in fasting, 30, 60, 90, and 120 minutes
Protein expression | 4 months (RCT) and 5 hours (crossover)
  Muscle sample assessed by means of western blotting
Gene expression | 4 months (RCT) and 5 hours (crossover)
  Muscle sample assessed by means of real-time PCR

IPD SHARING:
Plan to Share IPD: No